CLINICAL TRIAL: NCT06222580
Title: Safety and Efficacy of Dual Menin and FLT3 Inhibition in Patients With Relapsed/Refractory FLT3- Mutated Acute Myeloid Leukemia Containing a Concurrent MLL-Rearrangement or NPM1 Mutation: A Phase I (Ph I) Study of SNDX-5613 + Gilteritinib
Brief Title: SNDX-5613 and Gilteritinib for the Treatment of Relapsed or Refractory FLT3-Mutated Acute Myeloid Leukemia and Concurrent MLL-Rearrangement or NPM1 Mutation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Uma Borate (Other)
Responsible Party: Sponsor-Investigator, Uma Borate, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-23199; NCI-2024-00036 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-01-16; First posted 2024-01-24 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Acute Myeloid Leukemia With FLT3/ITD Mutation; Acute Myeloid Leukemia With KMT2A Rearrangement; Acute Myeloid Leukemia With NPM1 Mutation; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Specimen Handling; Biopsy; gilteritinib; revumenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (SNDX-5613 and gilteritinib) (Experimental): Patients receive SNDX-5613 PO BID and gilteritinib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow biopsy and aspiration, and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Gilteritinib; Drug: Revumenib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration and biopsy
Drug: Gilteritinib — Given PO
  Other Names: ASP-2215; ASP2215
Drug: Revumenib — Given PO
  Other Names: Menin-Mixed Lineage Leukemia Protein-Protein Interaction Inhibitor SNDX-5613; Menin-MLL Inhibitor SNDX-5613; Menin-MLL Interaction Inhibitor SNDX-5613; SNDX 5613; SNDX-5613; SNDX5613

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of SNDX-5613 and gilteritinib for treating patients with acute myeloid leukemia that has come back after a period of improvement (relapsed) or that does not respond to treatment (refractory) and has a mutation in the FLT3 gene along with either a mutation in the NMP1 gene or a type of mutation called a rearrangement in the MLL gene. SNDX-5613 is in a class of medications called menin inhibitors. It works by blocking the action of mutated MLL and NMP1 proteins that signal cancer cells to multiply. Gilteritinib is in a class of medications called tyrosine kinase inhibitors. It works by blocking the action of mutated FLT3 proteins that signal cancer cells to multiply. Giving SNDX-5613 with gilteritinib may be safe, tolerable and/or effective in treating patients with relapsed/refractory FLT3 mutated acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety of revumenib (SNDX-5613) + gilteritinib.

SECONDARY OBJECTIVES:

I. To determine the preliminary efficacy of SNDX- 5613+ Gilteritinib.

EXPLORATORY OBJECTIVES:

I. To perform pharmacokinetic and pharmacodynamics assessments of the study drug combination.

OUTLINE: This is a dose-escalation study.

Patients receive SNDX-5613 orally (PO) twice per day (BID) and gilteritinib PO once per day (QD) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow biopsy and aspiration, and blood sample collection throughout the study.

After completion of study treatment patients are followed up at 30 days and then every 12 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study
* Age ≥ 18 years at the date of signing the informed consent form (ICF)
* Morphologically confirmed diagnosis of the following based on 2022 World Health Organization (WHO) classification:

  * Relapsed or Refractory Acute Myeloid Leukemia with the following:

    * Refractory disease classified as having received 2 cycles of intensive induction or 2 cycles of hypomethylating agent (HMA) + Venetoclax with persistent disease of ≥ 5% blasts in the bone marrow and/or reappearance of peripheral blasts
  * FLT-3 mutated disease of the ITD or TKD subtype, AND
  * NPM1 mutation, MLL gene rearrangement and any other mutation that has proven HOXA-MEIS1 overexpression (NUP98, UBTF-TD, MLL-PTD and any others that have supporting literature)
* Patients must be receiving itraconazole, ketoconazole, posaconazole, or voriconazole (strong CYP3A4 inhibitors) for antifungal prophylaxis for at least 24 hours prior to enrollment and while on SNDX-5613 treatment. Patients must not be receiving any other strong CYP3A4 inhibitors/inducers
* Not suitable for immediate myeloablative/intensive chemotherapy based on investigator assessment of age, comorbidities, local guidelines, institutional practice (any or all of these)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 × ULN (except in the setting of isolated Gilbert syndrome)
* Estimated Glomerular Filtration Rate (eGFR) ≥ 60 mL/min/1.73m^2 (estimation based on Modification of Diet in Renal Disease (MDRD) formula, by local laboratory)
* Adequate cardiac function defined as ejection fraction (EF) of ≥50% by echocardiogram or multigated acquisition (MUGA) scan
* Patient can communicate with the investigator and has the ability to comply with the requirements of the study procedures
* Participants of childbearing potential must agree to have a negative serum pregnancy test at screening and a negative serum or urine pregnancy test on the first day of study treatment
* Participants capable of impregnating others who are having intercourse with people of childbearing potential must agree to abstain from intercourse or have their partner use 2 forms of contraception from the screening visit until 90 days after the last dose of study treatment. They must also refrain from sperm donation from the screening visit until 90 days following the last dose of study treatment
* Must be able to swallow the study medications
* Any prior treatment-related toxicities resolved to ≤ grade 1 prior to enrollment, with the exception of ≤ grade 2 neuropathy or alopecia
* Patients are not currently receiving the following therapies or have discontinued therapy based on the time periods below:

  * Radiation Therapy: At least 60 days from prior total body irradiation (TBI), craniospinal radiation and/or ≥ 50% radiation of the pelvis, or at least 14 days from local palliative radiation therapy (small port)
  * Stem Cell Infusion: At least 60 days must have elapsed from hematopoietic stem cell transplant (HSCT) and at least 4 weeks must have elapsed from donor lymphocyte infusion (DLI)
  * Immunotherapy: At least 42 days since prior immunotherapy, including tumor vaccines and checkpoint inhibitors, and at least 21 days since receipt of chimeric antigen receptor therapy or other modified T cell therapy
  * Antileukemia Therapy***: At least 14 days, or 5 half-lives, whichever is shorter, since the completion of antileukemic therapy (for example, but not limited to, small molecule or cytotoxic/myelosuppressive therapy), with the following exceptions:
  * Wah-out can be shorter for patients with rapidly progressing disease as determined by the treating investigator
  * Hydroxyurea for cytoreduction can be initiated without restriction related to timing of study entry. Hydroxyurea can be continued concomitantly with SNDX-5613, with medical monitor approval. Patients may continue to receive prophylactic intrathecal chemotherapy at any time at the treating physician's discretion
  * Hematopoietic Growth Factors: At least 7 days since the completion of therapy with short-acting hematopoietic growth factors and 14 days with long-acting growth factors
  * Biologics (e.g., monoclonal antibody therapy): At least 90 days, or 5 half-lives, whichever is shorter, since the completion of therapy with an antineoplastic biologic agent
  * Steroids: At least 7 days since systemic glucocorticoid therapy, unless receiving physiologic dosing (equivalent to ≤10 mg prednisone daily for patients ≥ 18 years or ≤10 mg/m^2 /day for patients

    * Prior treatment with gilteritinib is allowed

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia
* Diagnosis of extra-medullary acute myeloid leukemia (AML) based on WHO 2022 classification or myeloid sarcoma
* Suspected central nervous system (CNS) involvement. Patients with history of cerebrospinal fluid (CSF) involvement must either have documented CSF clearance prior to treatment initiation or be receiving active treatment for CNS involvement
* Participants with prior malignancy, except:

  * Participants with history of adequately treated malignancy for which no anticancer systemic therapy (namely chemotherapy, radiotherapy or surgery) is ongoing or required during the course of the study
  * Participants who are receiving adjuvant therapy such as hormone therapy are eligible. However, participants who developed therapy related neoplasms are not eligible
* Previous known allergy/sensitivity to components of gilteritinib or SNDX-5613. Prior treatment with gilteritinib is allowed and does not exclude a patient
* Patient with known human immunodeficiency virus (HIV) or has active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV). HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial. For patients with evidence of chronic HBV infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Individuals with a history of HCV infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Fridericia's corrected QT interval (QTcF) > 450 msec at time of screening
* Clinically significant ventricular arrhythmia (e.g., ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
* Uncontrolled intercurrent illness including, but not limited to, unstable angina pectoris, serious cardiac arrhythmia, myocardial infarction within 2 months prior to enrollment, New York Heart Association (NYHA) Class III or IV heart failure
* Patients with uncontrolled infection will not be enrolled until infection is treated and under control per the principal investigator or their designee
* Any psychiatric illness that prevents patient from informed consent process
* Pregnant or breastfeeding at the time of enrollment
* Patient has a malabsorption syndrome or other condition that precludes an enteral route of administration
* Patient has history of a cardiovascular, endocrinologic, hepatic, immunologic metabolic, neurologic, psychiatric, pulmonary, renal disease, or any other condition that in the opinion of the investigator would adversely affect his/her participation in this study or interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of hematologic adverse events (AEs) | Up to 30 days after completion of study treatment
  Adverse events will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. The toxicity data captured will include type, frequency, grade, severity, timing of onset, duration and relationship to study drug. Frequency tables will be used to summarize the AE data, where the number of patients with different types of AE will be tabulated by toxicity grade, counting only the highest grade of a certain type of AE occurred to the same patient. All adverse events regardless of attribution as well as those treatment- related AEs will be summarized.
Incidence of non-hematologic adverse events | Up to 30 days after completion of study treatment
  Adverse events will be graded according to CTCAE v5.0. The toxicity data captured will include type, frequency, grade, severity, timing of onset, duration and relationship to study drug. Frequency tables will be used to summarize the AE data, where the number of patients with different types of AE will be tabulated by toxicity grade, counting only the highest grade of a certain type of AE occurred to the same patient. All adverse events regardless of attribution as well as those treatment- related AEs will be summarized.
Recommended phase 2 dose for drug combination | During cycle 1 (28 days)
  Will be determined based on the maximum tolerated dose in conjunction with pharmacokinetic and pharmacodynamic assessments.

SECONDARY OUTCOMES:
Composite Complete Response Rate (CRc) | Up to 2 years
  Will be calculated in the efficacy analysis population and reported along with two-sided 95% exact binomial confidence limits.
Overall Response Rate | Up to 2 years
Rate of CRc with Measurable Residual Disease Negativity | Up to 2 years
  will be calculated in the efficacy analysis population and reported along with two-sided 95% exact binomial confidence limits.
Duration of response | From the date of first response to the earliest documentation of progressive disease, relapsed disease, or death, up to 2 years
  Will be calculated among patients who achieve a response and estimated using the method of Kaplan-Meier.
Overall Survival | From date of treatment start to death due to all cause, up to 2 years
  Will be estimated using the method of Kaplan-Meier.
Event Free Survival | From start of treatment to confirmed progressive disease, confirmed morphological relapse from complete remission or complete remission with incomplete hematologic recovery, treatment failure after at least 6 cycles of treatment or death, up to 2 years
  Will be estimated using the method of Kaplan-Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Uma M Borate, MD, MS, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (3):
- United States (3):
  - UNC Hospitals, University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu